CLINICAL TRIAL: NCT05311215
Title: A Randomized, Double-Blind, Placebo-Controlled Single Ascending Dose Escalation Study to Assess the Safety, Pharmacokinetics and Efficacy of SL-1002 in Patients With Limb Spasticity
Brief Title: Phase II Study to Assess Safety, Pharmacokinetics and Efficacy of SL-1002 for Limb Spasticity
Acronym: RAISE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saol Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Saol 1002-01
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SL-1002 (Experimental): SL-1002 injectable solution, single dose
  Interventions: Drug: SL-1002
- Matching placebo (Placebo Comparator): Matching placebo injectable solution, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SL-1002 — SL-1002 injectable solution
  Arms: SL-1002
Drug: Placebo — Matching placebo injectable solution
  Arms: Matching placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled single ascending dose escalation study intended to assess the safety, pharmacokinetics and efficacy of single treatment of SL-1002 in patients with mild to severe limb spasticity. The study will enroll 4 cohorts of 8 patients per cohort for a total of 32 patients. Patients will be randomized to receive either SL-1002 or placebo in a 3:1 ratio. The study period will be up to 26 weeks inclusive of a screening period of up to 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Spasticity based on MAS of greater than or equal to 2 in the specified limbs and muscle groups.
2. Patients who are diagnosed with spasticity of cerebral or spinal origin that can be treated with chemo denervation of the approved cohort-specific nerves. Prior history of chemo denervation must align with Exclusion #3 and #5 as noted below.
3. Patients who have had spasticity for greater than 6 months and have not had a significant change in their spasticity during recent evaluations or changes in dosing of spasticity medication in the 2 weeks prior to the Screening visit.
4. Male or female patients between 18-80 years of age, with a Body Mass Index (BMI) of 18.0 to 29.9 kg/m2 and a total body weight of ≥50.0 kg for males and ≥45.5 kg for females.
5. Female patients who are not pregnant.
6. Female patients of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration:

   1. Intra-uterine contraceptive device placed at least 4 weeks prior to study drug administration;
   2. Male condom with intravaginally applied spermicide starting at least 21 days prior to study drug administration;
   3. Hormonal contraceptives starting at least 4 weeks prior to study drug administration must agree to use the same hormonal contraceptive throughout the study;
   4. Sterile male partner (vasectomized since at least 6 months);
7. Female patients of non-childbearing potential as defined below:

   1. Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause).
   2. Pre-menopausal females with one of the following:
   3. Documented tubal ligation
   4. Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion
   5. Hysterectomy
   6. Documented bilateral oophorectomy.
8. Patients who are mentally coherent and responsive to communication, instructional command and have the ability to communicate proactively as defined by a Mini Mental State Examination (MMSE) score of 18 or greater. Patients can be enrolled into the study with or without the assistance of a caregiver based upon Investigator discretion. Patients who are cognitively compromised will be required to have a legally authorized representative consent for the study on their behalf.
9. Patients who have a positive response to baseline screening of 2-8mL lidocaine 1% solution administration.
10. Patients with no prior history or significant trauma to the injected limbs.

Exclusion Criteria:

1. Muscle contractures of the targeted upper or lower limb joints or any challenge that causes severe restriction of range of motion of targeted joints. Contractures will be identified by the Investigator following the lidocaine block by assessing the response.
2. Patients with severe muscle atrophy in the targeted limbs.
3. Patients who have had long-term treatments to block nerves (alcohol, phenol, etc.) that will be targeted in the study within 1 year of the Screening visit.
4. Patients currently on intrathecal or oral baclofen therapy for spasticity who have not been on a stable dose regimen for at least 2 weeks prior to the Screening Visit or who would need to have significant dose adjustments at any time point during study participation.
5. Patients who have received any botulinum toxin in the targeted muscle groups for the nerve block treatment within 6 months of the Screening Visit. Note: patients will not be able to receive any botulinum toxin injections to the targeted muscle group from the Screening Visit to the End of Study visit.
6. Patients with bleeding disorders or who are being treated with anticoagulants.
7. Patients with severe hepatic or renal impairment that, in the judgement of the Principal Investigator, will preclude participation in the study.
8. Female patients who are pregnant or planning to become pregnant during the duration of the study.
9. Female patients who are breast-feeding.
10. Patients who are unable or unwilling to comply with the requirements of the protocol.
11. Patients taking any of the following concurrent medications/over-the counter products (refer to Appendix 7 for a list of applicable medications):

    1. Probenecid or other OAT3 inhibitors.
    2. Inhibitors of CYP2E1, such as disulfiram.
12. Patients with known allergies or hypersensitivity to phenol and/or lidocaine and/or their excipients.
13. Documented history or evidence of alcohol or drug abuse within 1 year of the Screening Visit.
14. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days of the Screening Visit, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
15. Patients with clinically significant ECG abnormalities or vital sign abnormalities at the Screening Visit. Patients with ECG or vital sign abnormalities deemed non-clinically significant or unlikely to result in clinical compromise by the Principal Investigator may be considered for study inclusion.
16. Patients with clinically significant laboratory results at the Screening Visit (as judged by the Principal Investigator).
17. Any condition, in the opinion of the Principal Investigator, that may pose a significant risk to the patient, confound the results of the study or interfere significantly with the patient's participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events (TEAEs) overall | time of study drug administration to end of study visit (day 168)
  TEAE timepoints will be observed from the time point of administration of total dose until end of study visit (day 168)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - TIRR Memorial Hermann Research Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin